CLINICAL TRIAL: NCT06500702
Title: A Parallel-group Treatment, Phase 2a, Multicenter, Randomized, Double-blind, Placebo-controlled Umbrella Study to Evaluate the Efficacy and Safety of Frexalimab, Brivekimig, and Rilzabrutinib in Participants Aged 16 to 75 Years With Primary Focal Segmental Glomerulosclerosis (FSGS) or Minimal Change Disease (MCD)
Brief Title: A Study to Evaluate the Efficacy and Safety of Frexalimab, Brivekimig, or Rilzabrutinib in Participants Aged 16 to 75 Years With Primary Focal Segmental Glomerulosclerosis or Minimal Change Disease
Acronym: RESULT
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ACT18064; 2024-511775-15 (Registry Identifier: CTIS); U1111-1301-2676 (Registry Identifier: WHO)
Record Dates: First submitted 2024-07-08; First posted 2024-07-15 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Focal Segmental Glomerulosclerosis; Glomerulonephritis Minimal Lesion
MeSH Terms: conditions — Glomerulosclerosis, Focal Segmental; Nephrosis, Lipoid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Frexalimab (Experimental): Frexalimab active dose
  Interventions: Drug: frexalimab
- Brivekimig (Experimental): Brivekimig active dose
  Interventions: Drug: brivekimig
- Rilzabrutinib (Experimental): Rilzabrutinib active dose
  Interventions: Drug: rilzabrutinib
- Placebo (Placebo Comparator): Matching placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: frexalimab — frexalimab treatment
  Arms: Frexalimab
Drug: brivekimig — brivekimig treatment
  Arms: Brivekimig
Drug: rilzabrutinib — rilzabrutinib treatment
  Arms: Rilzabrutinib
Drug: placebo — placebo treatment
  Arms: Placebo

SUMMARY:
This is a parallel, Phase 2a, double-blind, 6-arm study for the treatment of primary focal segmental glomerulosclerosis (FSGS) or primary minimal change disease (MCD).

The purpose of this study is to measure the change in proteinuria and its impact on the rates of remission of nephrotic syndrome with frexalimab, brivekimig, or rilzabrutinib compared with placebo in participants with primary FSGS or primary MCD aged 16 to 75 years.

Study details for each participant include:

The study duration will be up to 76 weeks. The treatment duration will be 24 weeks. There will be up to 18 visits.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy report indicative of primary FSGS or primary MCD, with supportive clinical presentation per Investigator's judgement.
* UPCR ≥3 g/g at screening, or ≥ 1.5 g/g in those with eGFR ≥ 60.
* eGFR ≥45 mL/min/1.73 m^2 at screening.
* Documented history of UPCR (or 24-hour urine protein) reduction by >40% in response to corticosteroid or other immunosuppressive therapy when pre-treatment UPCR was ≥3.5 g/g (or pre-treatment 24-hr urine protein was ≥3.5 g/day if 24-hour urine protein is used).
* ≤10 mg/day prednisone or equivalent and stable starting at least 1 week prior to randomization.
* For those on a RAAS inhibitor prior to screening, the dose must be stable ≥4 weeks prior to screening; starting RAAS inhibitors or changing the dose will not be allowed during the double-blind or OLE treatment period.
* For those on an SGLT2 inhibitor prior to screening, the dose must be stable ≥4 weeks prior to screening; starting SGLT2 inhibitor treatment or changing the dose will not be allowed during the double-blind or OLE treatment periods.
* Body weight within 45 to 120 kg (inclusive) at screening.

Exclusion Criteria:

* Genetic or secondary FSGS or MCD. Those with APOL1 risk alleles are eligible.
* Collapsing variant of FSGS.
* ESKD requiring dialysis or transplantation.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 16 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2024-12-19 (Actual); Primary Completion 2026-12-23 (Estimated); Study Completion 2028-02-16 (Estimated)

PRIMARY OUTCOMES:
Percent reduction in urine protein to creatinine ratio (UPCR) | From baseline to Week 12

SECONDARY OUTCOMES:
Percentage of participants achieving FSGS partial remission endpoint | At Week 12
  Defined as UPCR ≤1.5 g/g and >40 % reduction of UPCR from baseline
Percentage of participants achieving CR | At Week 12
  Defined as UPCR ≤0.3 g/g
Incidence of treatment-emergent adverse events, treatment-emergent serious adverse events (SAEs), treatment-emergent adverse events of special interest (AESIs) and IMP discontinuation due to TEAEs during the study | Treatment emergent period, up to Week 48
  TEAEs, including clinically significant changes in vital signs, electrocardiogram [ECG], and laboratory evaluation
Plasma concentrations of frexalimab and rilzabrutinib and serum concentrations of SAR442970 | Up to Week 48
Occurrence of anti-drug antibodies (ADAs) against frexalimab and SAR442970 | Up to Week 48

CONTACTS AND LOCATIONS:
Locations (63):
- United States (14):
  - Investigational Site Number: 8400007, Birmingham, Alabama
  - Investigational Site Number: 8400015, Orange, California
  - Investigational Site Number: 8400012, San Francisco, California
  - Investigational Site Number: 8400014, Chicago, Illinois
  - Investigational Site Number: 8400017, Hinsdale, Illinois
  - Investigational Site Number: 8400010, Ann Arbor, Michigan
  - Investigational Site Number: 8400019, Edina, Minnesota
  - Investigational Site Number: 8400018, Las Vegas, Nevada
  - Investigational Site Number: 8400028, Albuquerque, New Mexico
  - Investigational Site Number: 8400001, New York, New York
  - Investigational Site Number : 8400021, Chapel Hill, North Carolina
  - Investigational Site Number: 8400024, Dallas, Texas
  - Investigational Site Number : 8400005, El Paso, Texas
  - Investigational Site Number: 8400016, Houston, Texas
- Argentina (2):
  - Investigational Site Number : 0320001, Buenos Aires
  - Investigational Site Number : 0320002, Córdoba
- Australia (2):
  - Investigational Site Number : 0360003, Garran, Australian Capital Territory
  - Investigational Site Number : 0360001, Parkville, Victoria
- Brazil (2):
  - Investigational Site Number: 0760002, São Paulo
  - Investigational Site Number: 0760001, São Paulo
- Canada (3):
  - Investigational Site Number : 1240002, London, Ontario
  - Investigational Site Number : 1240001, Montreal, Quebec
  - Investigational Site Number : 1240006, Québec, Quebec
- Chile (2):
  - Investigational Site Number : 1520003, Temuco, La Araucanía
  - Investigational Site Number : 1520002, Santiago, Reg Metropolitana de Santiago
- China (3):
  - Investigational Site Number : 1560001, Beijing
  - Investigational Site Number : 1560003, Chengdu
  - Investigational Site Number : 1560004, Shanghai
- Czechia (2):
  - Investigational Site Number : 2030002, Olomouc
  - Investigational Site Number : 2030001, Prague
- France (2):
  - Investigational Site Number : 2500002, Créteil
  - Investigational Site Number : 2500001, Paris
- Germany (2):
  - Investigational Site Number : 2760002, Berlin
  - Investigational Site Number : 2760003, Hanover
- Greece (3):
  - Investigational Site Number : 3000002, Athens
  - Investigational Site Number : 3000001, Heraklion
  - Investigational Site Number : 3000003, Ioannina
- Investigational Site Number : 3480001, Budapest, Hungary
- Italy (3):
  - Investigational Site Number : 3800002, Florence, Firenze
  - Investigational Site Number : 3800003, Naples, Napoli
  - Investigational Site Number : 3800001, Brescia
- Mexico (2):
  - Investigational Site Number : 4840001, Mexico City, Mexico City
  - Investigational Site Number : 4840003, Monterrey, Nuevo León
- Investigational Site Number : 5280001, Amsterdam, Netherlands
- Poland (2):
  - Investigational Site Number : 6160001, Lodz, Lódzkie
  - Investigational Site Number : 6160002, Opole, Opole Voivodeship
- Portugal (2):
  - Investigational Site Number : 6200001, Matosinhos Municipality
  - Investigational Site Number : 6200002, Porto
- Slovakia (3):
  - Investigational Site Number : 7030003, Banská Bystrica
  - Investigational Site Number : 7030004, Bratislava
  - Investigational Site Number : 7030001, Martin
- Spain (5):
  - Investigational Site Number : 7240001, Barcelona, Barcelona [Barcelona]
  - Investigational Site Number : 7240004, Barcelona, Catalunya [Cataluña]
  - Investigational Site Number : 7240005, Seville, Sevilla
  - Investigational Site Number : 7240002, Córdoba
  - Investigational Site Number : 7240003, Valencia
- Taiwan (2):
  - Investigational Site Number : 1580001, Taichung
  - Investigational Site Number : 1580002, Taipei
- Turkey (Türkiye) (2):
  - Investigational Site Number : 7920001, İzmit
  - Investigational Site Number : 7920002, Kayseri
- United Kingdom (3):
  - Investigational Site Number : 8260001, Leicester, Leicestershire
  - Investigational Site Number : 8260004, Salford, Manchester
  - Investigational Site Number : 8260005, Oxford, Oxfordshire

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- [Derived] Lin J, Radhakrishnan J. What Are Baskets, Umbrellas, and Platforms Doing in Nephrology Clinical Trials? J Am Soc Nephrol. 2025 Feb 3;36(8):1652-1654. doi: 10.1681/ASN.0000000648. No abstract available. PMID 39899371
- See also: ACT18064 Plain Language Results Summary — https://sanofi.trialsummaries.com/Study/StudyDetails?id=26033&tenant=MT_SNY_9011